CLINICAL TRIAL: NCT03155594
Title: Continuous Glucose Monitoring in the Hospital to Aid in Care and Improve Transition of Care to Outpatient
Brief Title: CGM to Aid Transition From Inpatient to Outpatient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Methodist Medical Center of Illinois (Other)
Responsible Party: Principal Investigator, Anne Webster, APN, APN, Methodist Medical Center of Illinois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1023056-2
Record Dates: First submitted 2017-05-09; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Diabete Mellitus
Keywords: Diabetes; Diabetes Mellitus; Diabetes Type 1; Diabetes Type 2; CGM; Continuous Glucose Monitoring; Inpatient; Outpatient; Transition of care; DM-1; DM-2; Freestyle Libre
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Adult patients in the hospital receiving 4-5 glucometer checks per day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm (Experimental): Patients in this trial will receive a FreeStyle Libre patch that continuously measures glucose in addition to their standard glucose monitoring.
  Interventions: Device: Freestyle Libre

INTERVENTIONS:
Device: Freestyle Libre — Continuous glucose monitoring patch

SUMMARY:
A pilot study using the FreeStyle Libre to assess its potential benefits in patients with diabetes starting when they are inpatients and continuing during the transition of care to the outpatient setting to see if diabetes care can be improved after discharge.

This study is designed to address the following questions:

1. How do the glucose readings from FreeStyle Libre Pro compare to our inpatient glucometer system? Is the system is accurate enough to use for clinical decision making?
2. How often does the additional continuous glucose data change inpatient care?
3. Does this technology work with inpatient nursing workflow?
4. Does leaving the patch on at discharge and reading in the office improve transition of care?
5. Does reading the patch after discharge in the office improve follow-up care?

DETAILED DESCRIPTION:
Continuous glucose monitoring checks blood glucose continuously. This allows the patient and provider to see what the glucose does between finger stick measurements. The FreeStyle Libre, is a sensor patch that can continuously measure glucose for up to two weeks.

Objectives To see if new continuous glucose technology can 1) Improve glucose management in the hospital compared to finger sticks 4-5 times per day. 2) Help with glucose control during transition of care from hospital to home and follow-up in the office The main hypothesis of this study is if the additional glucose information improves diabetes care for patients in the hospital and after the transition to home.

Background The FreeStyle Libre Pro was recently approved by the FDA. It is a patch applied to the skin with glucose containing sensing technology that will record the subcutaneous blood continuously for up to 2 weeks. It has the potential to reduce the number of painful glucose checks done by pricking the finger. It is currently approved for use in the office.

Study Method A pilot using the FreeStyle Libre to assess its potential benefits in patients with diabetes starting when they are inpatients and continuing during the transition of care to the outpatient setting to see if diabetes care can be improved after discharge. To our knowledge, there are currently no studies on using CGM to help the transition of care.

Protocol Outline

1. Apply the FreeStyle Libre Pro to patients in the on 4-5 glucose checks per day by finger stick with insulin ordered at least 4 times per day with patient consent.
2. Download the FreeStyle Libre each day and evaluate if the continuous data changes the treatment in the hospital.
3. The patient will continue to wear the patch on discharge to home.
4. At an after hospital office visit, the patient's data will again be downloaded and compared to finger stick glucoses done at home. Another evaluation well be done to see if this additional information changes therapy.
5. Additionally, an overall evaluation will be done comparing the glucoses on the FreeStyle Libre Pro with finger stick glucoses to evaluate if the accuracy is adequate for clinical decision making.

Population Studied Estimated number of subjects: 15 Age (inclusive) Ages 18 and above Sex (estimate M:F ratio) No sexual preference The population is patients in the hospital requiring 4-5 finger stick glucoses a day and orders on insulin. Patient should also be able to follow-up in the Diabetes Clinic to download and review the information and have no contraindication to the patch such as an adhesive allergy.

Recruitment Patient consulted for diabetes management in the hospital who are on 4-5 finger stick glucoses per day and insulin will be approached.

Risks and Benefits Benefits are chance to try new method of checking blood glucose. There are potential benefits if additional information improves their care. Downloads will be reviewed and shared with patients whenever possible. Risks are pain on application of the patch and possible allergies to the adhesive. (2) others: Potential benefit is improvement in diabetes care during hospitalization and transition of care. See no downside for others.

Alternative Treatments Standard care will be provided to all patients. They are under no obligation to try the patch. The patient may discontinue the patch and drop out of the study at any time. If the patient elects to enroll in the study, information from the patch download may be used to modify the treatment. If and how often this happens is one of the study outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients on insulin therapy 18 years and older on insulin with glucose testing 4-5 times per day
2. Patient able to sign informed consent.

Exclusion Criteria:

1. Patient unable to give informed consent
2. Critically ill patients will not be started in the CGM patch, but he patch will not be removed if transferred to ICU.
3. Patients currently on acetaminophen
4. Currently on diathermy treatments
5. Pregnancy
6. Dialysis
7. Currently on vitamin C
8. Patient is sensitive to the adhesive or develops significant skin irritation.
9. Treatment for dehydration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-07-15 (Estimated); Study Completion 2017-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in care | 2 weeks
  Each day a clinician from the Diabetes Service sees a patient in the hospital or office setting after discharge, they will download the information in the sensor patch. The clinician will note on the data collection sheet if the additional information changed the care compared to the information available from the hospital and patient glucose testing.

SECONDARY OUTCOMES:
Accuracy of device | 2 weeks
  Each glucometer glucose and serum glucose will be compared to the readings from the sensor patch.

CONTACTS AND LOCATIONS:
Overall Officials: David E. Trachtenbarg, MD, Study Chair — Methodist Medical Center of Illinois
Locations (1):
- Methodist Medica Center of Illinois, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beck RW, Riddlesworth T, Ruedy K, Ahmann A, Bergenstal R, Haller S, Kollman C, Kruger D, McGill JB, Polonsky W, Toschi E, Wolpert H, Price D; DIAMOND Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Adults With Type 1 Diabetes Using Insulin Injections: The DIAMOND Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):371-378. doi: 10.1001/jama.2016.19975. PMID 28118453
- [Background] Bailey KJ, Little JP, Jung ME. Self-Monitoring Using Continuous Glucose Monitors with Real-Time Feedback Improves Exercise Adherence in Individuals with Impaired Blood Glucose: A Pilot Study. Diabetes Technol Ther. 2016 Mar;18(3):185-93. doi: 10.1089/dia.2015.0285. Epub 2016 Feb 17. PMID 26885934
- [Background] Sato J, Kanazawa A, Ikeda F, Shigihara N, Kawaguchi M, Komiya K, Uchida T, Ogihara T, Mita T, Shimizu T, Fujitani Y, Watada H. Effect of treatment guidance using a retrospective continuous glucose monitoring system on glycaemic control in outpatients with type 2 diabetes mellitus: A randomized controlled trial. J Int Med Res. 2016 Feb;44(1):109-21. doi: 10.1177/0300060515600190. Epub 2015 Dec 7. PMID 26647072
- [Background] De Block CE, Gios J, Verheyen N, Manuel-y-Keenoy B, Rogiers P, Jorens PG, Scuffi C, Van Gaal LF. Randomized Evaluation of Glycemic Control in the Medical Intensive Care Unit Using Real-Time Continuous Glucose Monitoring (REGIMEN Trial). Diabetes Technol Ther. 2015 Dec;17(12):889-98. doi: 10.1089/dia.2015.0151. Epub 2015 Aug 25. PMID 26305390
- [Background] Schaupp L, Donsa K, Neubauer KM, Mader JK, Aberer F, Holl B, Spat S, Augustin T, Beck P, Pieber TR, Plank J. Taking a Closer Look--Continuous Glucose Monitoring in Non-Critically Ill Hospitalized Patients with Type 2 Diabetes Mellitus Under Basal-Bolus Insulin Therapy. Diabetes Technol Ther. 2015 Sep;17(9):611-8. doi: 10.1089/dia.2014.0343. Epub 2015 Apr 30. PMID 25927357
- [Background] Kusunoki Y, Katsuno T, Nakae R, Watanabe K, Akagami T, Ochi F, Tokuda M, Murai K, Miuchi M, Miyagawa J, Namba M. Evaluation of blood glucose fluctuation in Japanese patients with type 1 diabetes mellitus by self-monitoring of blood glucose and continuous glucose monitoring. Diabetes Res Clin Pract. 2015 May;108(2):342-9. doi: 10.1016/j.diabres.2015.01.040. Epub 2015 Mar 4. PMID 25779865
- [Background] Joubert M, Fourmy C, Henri P, Ficheux M, Lobbedez T, Reznik Y. Effectiveness of continuous glucose monitoring in dialysis patients with diabetes: the DIALYDIAB pilot study. Diabetes Res Clin Pract. 2015 Mar;107(3):348-54. doi: 10.1016/j.diabres.2015.01.026. Epub 2015 Jan 21. PMID 25638452
- [Background] Kepenekian L, Smagala A, Meyer L, Imhoff O, Alenabi F, Serb L, Fleury D, Dorey F, Krummel T, Le Floch JP, Chantrel F, Kessler L. Continuous glucose monitoring in hemodialyzed patients with type 2 diabetes: a multicenter pilot study. Clin Nephrol. 2014 Oct;82(4):240-6. doi: 10.5414/CN108280. PMID 25161114
- [Background] Boom DT, Sechterberger MK, Rijkenberg S, Kreder S, Bosman RJ, Wester JP, van Stijn I, DeVries JH, van der Voort PH. Insulin treatment guided by subcutaneous continuous glucose monitoring compared to frequent point-of-care measurement in critically ill patients: a randomized controlled trial. Crit Care. 2014 Aug 20;18(4):453. doi: 10.1186/s13054-014-0453-9. PMID 25139609
- See also: Device website — http://www.freestylelibrepro.us/index.html